CLINICAL TRIAL: NCT01680211
Title: Efficacy and Safety Study of Herbal Supplements (SR-L-01, SR-B-01 and SI-S-01) in the Management of Prediabetes and Mild to Moderate Hyperlipidemia
Brief Title: Safety and Efficacy Study of Herbal Supplements in Prediabetic and Mild to Moderate Hyperlipidemic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olive Lifesciences Pvt Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OL-S-OB-LP/03-12; CTRI/2012/05/002678 (Registry Identifier: Clinical Trials Registry - India (CTRI))
Record Dates: First submitted 2012-08-29; First posted 2012-09-07 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Prediabetes; Hyperlipidemia
Keywords: Blood Sugar,; Lipoproteins,; Salacia,; Sesame,; Prediabetes,; Hyperlipidemia,; Herbal supplement
MeSH Terms: conditions — Prediabetic State; Hyperlipidemias; SeSAME syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Salacia bark extract (SR-B-01) and TLC (Experimental): Capsules containing 250mg of salacia bark extract,two times a day along with Therapeutic Lifestyle Change (TLC)
  Interventions: Dietary Supplement: Salacia bark extract; Behavioral: TLC
- Sesame seeds extract (SI-S-01) and TLC (Experimental): Capsules containing 250mg of sesame seed extract,two times a day along with Therapeutic Lifestyle Change (TLC)
  Interventions: Dietary Supplement: Sesame seed extract; Behavioral: TLC
- Salacia leaf extract (SR-L-01) and TLC (Experimental): Capsules containing 250mg of salacia leaf extract,two times a day along with Therapeutic Lifestyle Change (TLC)
  Interventions: Dietary Supplement: Salacia leaf extract; Behavioral: TLC
- Placebo and TLC (Placebo Comparator): Capsules containing 250mg of placebo,two times a day along with Therapeutic Lifestyle Change (TLC)
  Interventions: Behavioral: TLC; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Salacia bark extract
  Arms: Salacia bark extract (SR-B-01) and TLC
Dietary Supplement: Salacia leaf extract
  Arms: Salacia leaf extract (SR-L-01) and TLC
Dietary Supplement: Sesame seed extract
  Arms: Sesame seeds extract (SI-S-01) and TLC
Behavioral: TLC — Lifestyle changes include diet, exercise, weight loss, etc.
Other: Placebo
  Arms: Placebo and TLC

SUMMARY:
Objective of this study is to determine the safety and efficacy of administration of herbal supplements (Salacia leaf extract, Salacia root extract and Sesame seed extract) for 6 weeks in the management of prediabetes and mild to moderate hyperlipidemia.

ELIGIBILITY:
Inclusion Criteria:

1. As per ATP III guidelines: Baseline LDL ranging 160-189 mg/dL, TC >200 mg/dL and with no or one of the below risk factors

   * Current cigarette smoking
   * Family history of premature Coronary Heart Disease(CHD); in male first degree relative <55 years; in female first degree relative <65 years)
   * Hypertension (BP >140/90 mmHg or on antihypertensive medication)
   * Low HDL-C (<40 mg/dL)
   * Age (men > 40 years)
2. Impaired glucose tolerance (2-hour post 75 g OGTT glucose levels in the range of ≥140 to ≤ 200 mg/dL)
3. Impaired fasting sugar (Fasting blood sugar levels in the range of ≥ 100 to ≤125 mg/dL)
4. Being mentally competent and able to understand all study requirements and sign the informed consent form.

Exclusion Criteria:

1. Patients with severe liver, renal, cardiac or brain diseases.
2. Pregnant or lactating women or women of child bearing potential whom are not practicing a reliable form of birth control (either with IUD or with stable usage of oral contraceptives).
3. Unable to complete follow up.
4. Subjects on any medication that would affect evaluation like Statins.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in Blood Sugar and lipid profiles | baseline and 6 weeks
  Change in of blood sugar out come will be measured by Fasting Blood Sugar (FBS), Oral Glucose Tolerance Test (OGTT) and Postprandial Blood Sugar (PPBS). Change in lipid profiles are measured by Low Density Lipoprotein (LDL), Very Low Density Lipoprotein (VLDL), High Density Lipoprotein (HDL) and Total Cholesterol (TC).

SECONDARY OUTCOMES:
Clinical laboratory evaluations | 0 and week 6
  Electrocardiography (ECG), haematology (Complete Blood Count), biochemical tests (blood urea, and serum creatinine), liver function tests and urine routine analysis

CONTACTS AND LOCATIONS:
Overall Officials: K R Raveendra, M.D, Principal Investigator — Srinivasa Clinic & Diabetic Care Center
Locations (1):
- Srinivasa Clinic & Diabetic Care Center, Bangalore, Karnataka, India